CLINICAL TRIAL: NCT05696405
Title: Thoracoscopic Treatment of Mediastinal Ectopic Parathyroid Adenomas: A Case Series and Literature Review
Brief Title: VATS for Resection of Mediastinal Parathyroids
Status: Completed | Type: Observational
Sponsor: Hospital General Ajusco Medio (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Karla Verónica Chavez-Tostado, MD, Hospital Reg. Lic. Adolfo Lopez Mateos
Other Study IDs: 004
Record Dates: First submitted 2023-01-12; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Mediastinal Parathyroid Adenoma; Hyperparathyroidism
Keywords: hyperparathyroidism; Video-assisted thoracoscopy surgery; Mediastinal ectopic parathyroid adenoma
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: VATS resection of MEPA — VATS resection of mediastinal parathyroid adenoma

SUMMARY:
Background: hyperparathyroidism (HPT) is a disease caused by hypersecretion of one or more parathyroid glands, it can be associated with ectopic mediastinal parathyroid glands (MEPA) in 2% of cases. The use of video-assisted thoracoscopic surgery (VATS) for the surgical resection of these glands is a safe, cost-effective, and low-morbidity option for patients with MEPA. We report a case series of patients with this disease managed with VATS.

Patients & Methods: From 2008 to 2022, a retrospective study involving patients with MEPA and treated by VATS approach was performed in a tertiary hospital in Mexico City. Relevant biochemical and clinical variables such as imaging studies, pre and postoperative lab results, surgical strategy and outcomes, and pathological analyses were analyzed.

DETAILED DESCRIPTION:
Hyperparathyroidism (HPT) is a clinical disorder characterized by an inappropriately elevated paratohormone (PTH) due to hypersecretion of one or more parathyroid glands, that may develop secondary hypercalcemia and other metabolic disturbances. This disease includes various signs and symptoms such as nephrolithiasis, osteopenia and osteoporosis, depression, mental numbness, loss of appetite, nausea, vomiting, constipation among others. The abnormal secretion of PTH is most commonly caused by a single parathyroid gland adenoma in 85% of the cases, in the other 15% is due to multiple gland hyperplasia (15-20%)(1) or rarely from a parathyroid carcinoma (<1%). HPT occurs in both genders equally around the sixth decade(2). World HPT prevalence is estimated at 1 in every 500 women and 1 in every 2000 men(3).

Mediastinal ectopic parathyroid adenomas (MEPA) are rare tumors, constituting 1-2% of all parathyroid adenomas. These glands are inferior to the sternal notch and their location may vary from the superior mediastinum to the pericardium and diaphragm(4). The first report of a mediastinal parathyroid adenoma was in 1932 by Churchill in the patient Captain Charles E. Martell, who had 6 prior cervical explorations for his hyperparathyroidism until an ectopic gland was found in the superior mediastinum(5). Before the introduction of VATS, MEPA were usually resected by thoracotomy or a median sternotomy, currently with the daily use of minimally invasive surgery, VATS is being adopted as the procedure of choice.

The aim of this study to report a case series of patients with MEPA treated with VATS, along with a literature review.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MEPA

Exclusion Criteria:

* incomplete records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with MEPA and treated by VATS approach was performed in a tertiary hospital in Mexico City.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Biochemical cure of hyperparathyroidism | 24hours
  Normalization of Paratohormone leves

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kitada M, Yasuda S, Nana T, Ishibashi K, Hayashi S, Okazaki S. Surgical treatment for mediastinal parathyroid adenoma causing primary hyperparathyroidism. J Cardiothorac Surg. 2016 Apr 7;11:44. doi: 10.1186/s13019-016-0461-8. PMID 27056365
- [Result] Long KL, Lee CY, Ramaiah C, Sloan DA. Intrapericardial parathyroid adenomadagger. J Surg Case Rep. 2013 Aug 29;2013(8):rjt064. doi: 10.1093/jscr/rjt064. PMID 24964470
- [Result] Hu J, Ngiam KY, Parameswaran R. Mediastinal parathyroid adenomas and their surgical implications. Ann R Coll Surg Engl. 2015 May;97(4):259-61. doi: 10.1308/003588415X14181254789088. PMID 26263931
- [Result] Spence HM. The life and death of Captain Charles Martell and kidney stone disease. J Urol. 1984 Dec;132(6):1204-7. doi: 10.1016/s0022-5347(17)50098-1. PMID 6389906
- [Result] Sreevathsa MR, Melanta K. Unilateral Exploration for Parathyroid Adenoma. Indian J Surg Oncol. 2017 Jun;8(2):142-145. doi: 10.1007/s13193-016-0605-2. Epub 2016 Dec 27. PMID 28546708
- [Result] Wilhelm SM, Wang TS, Ruan DT, Lee JA, Asa SL, Duh QY, Doherty GM, Herrera MF, Pasieka JL, Perrier ND, Silverberg SJ, Solorzano CC, Sturgeon C, Tublin ME, Udelsman R, Carty SE. The American Association of Endocrine Surgeons Guidelines for Definitive Management of Primary Hyperparathyroidism. JAMA Surg. 2016 Oct 1;151(10):959-968. doi: 10.1001/jamasurg.2016.2310. PMID 27532368
- [Result] Medrano C, Hazelrigg SR, Landreneau RJ, Boley TM, Shawgo T, Grasch A. Thoracoscopic resection of ectopic parathyroid glands. Ann Thorac Surg. 2000 Jan;69(1):221-3. doi: 10.1016/s0003-4975(99)01127-3. PMID 10654517